CLINICAL TRIAL: NCT03047577
Title: Brief Intervention for ICU Patients with Alcohol Use Disorders- a Randomized Controlled Trial
Brief Title: Brief Intervention for ICU Patients with Alcohol Use Disorders
Acronym: ICU-BI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting stopped due to slow recruitment particularly due to COVID
Sponsor: University of Helsinki (Other)
Collaborators: Tampere University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Johanna Hastbacka, Dr, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYH2017105
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Use Disorder; Critically Ill
Keywords: Brief intervention; Alcohol; Alcohol use disorder; Intensive care unit; Critically ill; Audit
MeSH Terms: conditions — Alcoholism; Critical Illness | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to a standard care or an intervention arm
Who Masked: Outcomes Assessor
Masking Description: Unlike other team members, the investigator interviewing the patients will be unaware of the treatment group. The patient will be encouraged not to reveal the treatment group to the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care arm (No Intervention): Treatment as usual and discussion according to the treating clinicians in the hospital
- Intervention arm (Other): Patients receive a brief intervention, including a short discussion, opportunity for an appointment with a social worker and written information about effects of alcohol on health and contact information for seeking additional support
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — A 15-20minute discussion about the patients alcohol use and its association with current health conditions, option for a discussion with social worker and written material (information about how alcohol affects health and contact details for seeking more support)
  Other Names: Mini-intervention
  Arms: Intervention arm

SUMMARY:
Patients non-electively admitted to intensive care units (ICUs) will be screened for eligibility. The investigators will include adult patients with risk level alcohol use, defined by AUDIT-C score (>5 for females, >6 for males). Informed consent will be obtained from the patient in the end or shortly after the ICU treatment, when they have regained sufficient cognitive function. 600 patients will be randomized to receive either routine treatment or a brief intervention (BI). The BI includes a 20 minute discussion with pre-educated study personnel, option to discussion with a social worker and written material. Primary outcome measure is the amount of alcohol used during the preceding week (g/week), at 6 and 12 months after study entry. The information will be obtained 1)in an interview by a study team member blinded for the intervention arm at 6 months 2) A letter of a telephone interview at 12 months. AUDIT score, EQ-5D and mortality will also be recorded.

An interim analysis by an external reviewer will be performed after the primary outcome has been recorded for 200 patients,

ELIGIBILITY:
Inclusion Criteria:

* AUDIT-C score >5 (women) and >6 (men)
* Non-elective admission to the ICU

Exclusion Criteria:

* Terminal illness (expected to survive less than 6 months), palliative care
* Diagnosed severe mental illness (psychos, severe depression, bipolar disorder, personality disorder)
* Cognitive disability
* Diagnosed dementia
* Impaired level of consciousness at discharge from the ICU (expected to remain unchanged >2 days
* Other substance abuse (excluding cigarette smoking)
* Ongoing treatment for alcohol dependency
* Insufficient language skills (finnish/swedish)
* Expected difficulty in getting contacted by mail or telephone (no permanent address or telephone in use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Reported total amount of alcohol consumed during preceding week | 6 months after study enrollment
  The patients are interviewed and the amount of alcohol consumed during the last week is recorded and converted in grams
Reported total amount of alcohol consumed during preceding week | 12 months after study enrollment
  The patients are interviewed and the amount of alcohol consumed during the last week is recorded and converted in grams

SECONDARY OUTCOMES:
Change in AUDIT score | 6 months after study enrollment
  The AUDIT score will be filled in an interview and compared with the initial score obtained on study admission
Change in AUDIT score | 12 months after study enrollment
  The AUDIT score will be filled in a telephone interview or by mailed questionnaire and compared with the initial score obtained on study admission
Mortality | One year after study enrollment
  Survival of the patients will be obtained from Statistics Finland
Quality of life | One year after study enrollment
  A structured questionnaire EQ-5D will be mailed or filled in a telephone interview and the EQ-5D will be compared between the groups

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Helsinki University Hospital Intensive Care Units 20 and M1, Helsinki, Helsinki
  - Tampere University Hospital ICU, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nissila E, Hynninen M, Jalkanen V, Kuitunen A, Backlund M, Inkinen O, Hastbacka J. The effectiveness of a brief intervention for intensive care unit patients with hazardous alcohol use: a randomized controlled trial. Crit Care. 2024 Apr 30;28(1):145. doi: 10.1186/s13054-024-04925-z. PMID 38689346